CLINICAL TRIAL: NCT03816501
Title: The Effect of Favorite Music on Postoperative Anxiety and Pain
Brief Title: Effect of Preoperative Music on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Kavak Akelma, anesthesiology and reanimation specialist doctor, Ankara Diskapi Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Anxiety
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Music on Postoperative Anxiety
Keywords: postoperative anxiety; State - Trait Anxiety Inventory
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music (Other): The preference of the patients will be listened to preoperatively through the headphones.
  Interventions: Other: music
- no music (Other): preoperative music will not be listened
  Interventions: Other: no music

INTERVENTIONS:
Other: music — The preference of the patients will be listened to preoperatively through the headphones
  Arms: music
Other: no music — the patients will not be listened
  Arms: no music

SUMMARY:
In this study, we are planning to evaluate whether listening to the music of the patient's choice preoperatively contributes to postoperative anxiety.

DETAILED DESCRIPTION:
Preoperative anxiety can be detected via structured and standardised screening by the State - Trait Anxiety Inventory (STAI) I and II.

117 patients scheduled for inguinal hernia surgery for any reason in the age range of 18-70 will be included in our study. preoperative STAI I and II score (anxiety questionnaire) will be applied to each patient. The patients will be divided into two groups as preoperative music played and not played. The list of patients listening to the music will be played through the headphones which are the preference of the patients. The postoperative STAI questionnaire will be applied again. results will be evaluated statistically

ELIGIBILITY:
Inclusion Criteria:

* inguinal hernia surgery
* speak Turkish language

Exclusion Criteria:

* Patients with dementia and psychiatric disorders
* anxiolytic and psychiatric drug users
* patients without written consent
* poor vision,
* significant hearing loss,
* active opioid use,
* unwillingness to participate in the study
* unwillingness to listening to music

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
STAI score | 24 hours
  preoperative and postoperative STAI I and II score questions will be asked.
11-point numerical rating scale (NRS) | 24 hours
  11-point numerical rating scale for pain (0='no pain' and 10='worst pain possible pain') were explained.

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Teaching and Research Hospital, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No